CLINICAL TRIAL: NCT04015063
Title: A Single-Arm, Open-Label, Single Center Clinical Study to Evaluate the Efficacy and Safety of P29429-01 in Aging Facial Skin
Brief Title: Efficacy and Safety of Skin Care Product in Aging Facial Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201810063RSD
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2018-12

CONDITIONS: Skin Aging
Keywords: Dermatology; Skin Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Subjects (Other): Women subjects 40-65 years of age that meet the specified inclusion/exclusion criteria taking P29429-01 as a skin care product per the protocol.
  Interventions: Other: Anti-Aging Skin Care product

INTERVENTIONS:
Other: Anti-Aging Skin Care product — Primary Subjects will use P29429-01 as an anti-aging skin care product on full face twice a day for 12-week.
  Other Names: P29429-01

SUMMARY:
The purpose of this study is to assess the efficacy and safety of P29429-01 as a skin care product to manage skin aging in women subjects 40-65 years of age.

DETAILED DESCRIPTION:
Background and Rationale:

Skin aging, a major concern for females, is closely associated with factors including genetics, age and UV exposure.

Its first signs include reduced epidermal and dermal thickness, reduced water content in the stratum corneum causing the "dry look" of skin.

The ability of dermal fibroblasts to synthesize collagen fibers is reduced bring the decreased collagen content, and the intradermal elastic fibers are denatured and lose elasticity. The extracellular matrix of the dermis, such as hyaluronic acid, are also decreasing year by year.

These are the primary causes of wrinkle formation, loosening and drooping. The anti-aging product used in this study, P29429-01, is developed and manufactured by Orient EuroPharma. Its main ingredients include Hesperetin, a citrus bioflavonoid of antioxidant activity extracted from citrus peel. It is widely used in cosmetic products. Sodium cyclic lysophosphatidic acid, a substance extracted from soybean, increases hyaluronic acid and collagen synthesis in the skin to achieve hydration and anti-aging.

In this study, subjects are subject to a 4-week washout period before using P29429-01 on full face twice a day for 12-week. A skin analyzer is used to obtain skin aging indices to assess the efficacy and safety of P29429-01.

Study Purpose:

The purpose of this study is to assess the efficacy and safety of P29429-01 as a skin care product to manage skin aging in women subjects 40-65 years of age who show manifestations of facial skin aging. Subjects are to undergo a 4-week washout period before using P29429-01 on the face for 12 weeks. A skin analyzer is used to obtain skin aging indices for said assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Females 40~65 years of age;
2. Subjects are not found with facial skin tissue changes or inflammation as determined by the investigator ;
3. Has skin aging of Glogau class II, i.e. presence of wrinkles during facial movement or resting, as determined by the investigator;
4. The subject is able to understand and comply with the requirements, instructions and restrictions specified in the protocol; and
5. Sign on the informed consent form.

Exclusion Criteria:

1. Received active facial treatment including laser, pulse light, CPT Thermage, HIFU lifting or subcutaneous filler injection in the last 6 months;
2. Has history of chronic skin condition or autoimmune disorders such as atopic dermatitis, psoriasis, chronic urticaria, vitiligo, rosacea or keloid;
3. Has history of allergy to the study skin care product (P29429-01) compositions, moisturizer or sunscreen;
4. Pregnant or breastfeeding women;
5. Received hormone medications such as estrogen or progesterone, or health foods such as royal jelly, soybean isoflavone, red clover, black cohosh, Chinese Angelica, evening primrose oil, borage oil, chasteberry or placenta extract within 30 days before the study;
6. Required treatment for any acute condition or infection within 14 days before the study;
7. Experienced a serious medical condition such as disease of the heart, lungs, brain and/or liver within 3 months before the study;
8. Has been a routine smoker within 12 months before the study;
9. Currently has malignant tumor;
10. Has used any medicine for skin use on the face that is deemed to interfere with the study within 30 days before the study by investigator;
11. Has participated in another clinical trial within 30 days before the study;
12. Receiving medical management that may affect the ability to participate in this study;
13. Inappropriate for participating in this study as deemed by the principal investigator.

Inclusion Criteria for Substudy:

1. Has provided written informed consent for the main study;
2. Subjects are not found with tissue changes or inflammation at the planned biopsy site on medial forearm skin as determined by the principal investigator or dermatologist;
3. The subject is able to understand and comply with the requirements, instructions and restrictions specified in the substudy;
4. Sign and date on the informed consent form of the substudy.

Exclusion Criteria for Substudy:

1. Currently using anticoagulants;
2. Patients with severe coagulation disorder;
3. Patients with keloid predisposition.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-05 (Estimated); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
Facial skin hydration change from baseline | Week 12
  Corneum hydration of the skin will be determined using CK's Corneometry
Facial skin elasticity change from baseline | Week 12
  Elasticity of the skin will be determined using CK's Cutometer.

SECONDARY OUTCOMES:
Facial spots change from baseline | Week 12
  Assess facial skin spots with VISIA advanced skin tester.
Facial pores change from baseline | Week 12
  Assess pore size with VISIA advanced skin tester.
Facial wrinkles change from baseline | Week 12
  Assess wrinkles with VISIA advanced skin tester.
Facial texture change from baseline | Week 12
  Assess texture with VISIA advanced skin tester.
Facial porphyrin (from Propionibacterium acnes) change from baseline | Week 12
  Assess porphyrin values with VISIA advanced skin tester.
Facial brown spots change from baseline | Week 12
  Assess brown spots with VISIA advanced skin tester.
Facial red area change from baseline | Week 12
  Assess red area with VISIA advanced skin tester.
Facial UV spots change from baseline | Week 12
  Assess UV spots with VISIA advanced skin tester.
Sebumeter values change from baseline | Week 12
  Measure sebum (oil) on the skin with CK skin tester.
Mexameter values change from baseline | Week 12
  Measure melanin content on the skin with CK skin tester.
Transepidermal water loss (TEWL) by tewameter change from baseline | Week 12
  Transepidermal water loss (TEWL) with CK skin tester.
Facial skin wrinkles change from baseline | Week 12
  Obtain and assess wrinkles with Antera 3D tester.
Facial skin texture change from baseline | Week 12
  Obtain and assess texture with Antera 3D tester.
Facial skin pore change from baseline | Week 12
  Obtain and assess pore size with Antera 3D tester.
Facial skin depression/elevation change from baseline | Week 12
  Obtain and assess depression/elevation with Antera 3D tester.
Facial skin melanin values change from baseline | Week 12
  Obtain and assess melanin values with Antera 3D tester.
Facial skin hemoglobin values change from baseline | Week 12
  Obtain and assess hemoglobin values with Antera 3D tester.
Assess the safety of P29429-01 as a skin care product | Week 1~12
  Assess the incidence of adverse events.
Assess the safety of P29429-01 as a skin care product with skin health questionnaires | Week 1~12
  The skin health questionnaires is an ordinal scale used to assess the skin health, such as skin inflammation ,red, scaling, itchy, and achy.
Study compliance of the subjects | Week-4~12
  Assess with phone calls and clinic visits.
Assess P29429-01 satisfaction of the subjects with satisfaction questionnaires | Week 1~12
  The satisfaction questionnaires is a Likert scale used to assess satisfaction of the subjects, such as improvement of facial skin hydration, elasticity, wrinkles, texture and appearance.
The effect of P29429-01 in increasing hyaluronic acid, collagen and elastic fiber using skin tissue biopsy | At week -1 and Week 12
  For subjects agreeing to provide a skin tissue biopsy, the skin biopsy is obtained from a small area on the medial side of the forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hua Liao, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hosptal, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black MM. A modified radiographic method for measuring skin thickness. Br J Dermatol. 1969 Sep;81(9):661-6. doi: 10.1111/j.1365-2133.1969.tb16204.x. No abstract available. PMID 5361423
- [Background] Uitto J, Fazio MJ, Olsen DR. Molecular mechanisms of cutaneous aging. Age-associated connective tissue alterations in the dermis. J Am Acad Dermatol. 1989 Sep;21(3 Pt 2):614-22. PMID 2674224
- [Background] Melchini A, Catania S, Stancanelli R, Tommasini S, Costa C. Interaction of a functionalized complex of the flavonoid hesperetin with the AhR pathway and CYP1A1 expression: involvement in its protective effects against benzo[a]pyrene-induced oxidative stress in human skin. Cell Biol Toxicol. 2011 Oct;27(5):371-9. doi: 10.1007/s10565-011-9194-6. Epub 2011 Jul 1. PMID 21720915